CLINICAL TRIAL: NCT02127294
Title: Effectiveness and Safety of Transcatheter Patent Foramen Ovale Closure for Migraine
Acronym: EASTFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFO-1shsf
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Foramen Ovale, Patent; Migraine
Keywords: Foramen Ovale, Patent; migraine; transcatheter patent foramen ovale closure; contrast-enhanced transcranial Doppler; Transthoracic Echocardiography
MeSH Terms: conditions — Foramen Ovale, Patent; Migraine Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcatheter closure group (Experimental): Migraine patients with patent foreman ovale (PFO)，who meet the criteria and agree to conduct closure of patent foramen ovale will be selected to this group.
  Interventions: Device: transcatheter patent foreman ovale closure
- Contrast group (No Intervention): Migraine patients with PFO，who meet the criteria but don't agree to conduct closure of patent foramen ovale will be selected to this group.

INTERVENTIONS:
Device: transcatheter patent foreman ovale closure
  Arms: Transcatheter closure group

SUMMARY:
The purpose of the study is to evaluate effectiveness and safety of transcatheter patent foramen ovale closure for migraine.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of migraine diagnosed by a neurologist according to the International Classification of Headache Disorders
* Transcranial Doppler evidence of right-to-left shunt(RLS) and echocardiographic evidence of PFO，of which the degree is moderate to large RLS
* Subjects who have not responded to or cannot take common migraine preventive medications
* Willing to participate in follow-up visits

Additional Inclusion Criteria:

* Transcatheter closure group: Closure of PFO is performed
* Contrast group: Subjects who meet the Inclusion Criteria, but refuse to undergo closure procedure

Exclusion Criteria:

* Seizure disorder
* Other organic central nervous system disease
* Subjects whose headaches are other than migraine, such as a result of traumatic head or neck injury
* Evidence of alcohol, drug or substance abuse within the previous year

Additional Exclusion Criteria for Transcatheter closure group:

* Subjects with intracardiac thrombus or tumor
* Subjects who have an acute or recent (within 6 months) myocardial infarction or unstable angina
* Subjects with left ventricular aneurysm or akinesis
* Subjects with atrial fibrillation/atrial flutter (chronic or intermittent)
* Subjects with another source of right to left shunt identified at baseline, including an atrial septal defect and/or fenestrated septum
* Subjects with contraindication to aspirin or Clopidogrel therapy
* Pregnant or desire to become pregnant within the next year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Contrast-enhanced Transcranial Doppler | within one year period
  Patients in transcatheter closure group are required to perform contrast-enhanced Transcranial Doppler at 1 month, 3 month, 6 month and 1 year after closure, respectively.

SECONDARY OUTCOMES:
Headache Impact Test-6 | within one year period, at least 3 months
  All patients complete HIT-6 score at baseline. Patients in transcatheter closure group follow-up at 1 month, 3 month, 6 month and 1 year after closure, respectively. Patients in contrast group follow-up twice during one year period.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, MD, PhD, Study Chair — The First Hospital of Jilin University; Yingqi Xing, MD, PhD, Study Director — The First Hospital of Jilin University; Yuzhu Guo, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Background] Yang Y, Guo ZN, Wu J, Jin H, Wang X, Xu J, Feng J, Xing Y. Prevalence and extent of right-to-left shunt in migraine: a survey of 217 Chinese patients. Eur J Neurol. 2012 Oct;19(10):1367-72. doi: 10.1111/j.1468-1331.2012.03793.x. Epub 2012 Jun 30. PMID 22747847
- [Derived] Xing YQ, Guo YZ, Gao YS, Guo ZN, Niu PP, Yang Y. Effectiveness and Safety of Transcatheter Patent Foramen Ovale Closure for Migraine (EASTFORM) Trial. Sci Rep. 2016 Dec 14;6:39081. doi: 10.1038/srep39081. PMID 27966652